CLINICAL TRIAL: NCT06806228
Title: Phase I Pilot Study to Evaluate the Anti-glioblastoma Effect of S-Gboxin in Standard Treatment of Glioblastoma/Diffuse Midline Glioma and Response to Treatment (Regardless of Mutation Status)
Status: Suspended | Phase: Phase 1 | Type: Interventional
Why Stopped: The study protocol will be changed
Sponsor: Petrov, Andrey (Other)
Collaborators: Lytvin,Ruslan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STM 0125-2G
Record Dates: First submitted 2025-01-26; First posted 2025-02-04 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Glioblastoma Multiforme; Diffuse Midline Glioma, H3 K27M-Mutant; Gliosarcoma; Giant Cell Glioblastoma; GBM
MeSH Terms: conditions — Glioblastoma; Gliosarcoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients will be offered 4 courses of Gboxin during (or without) standard treatment. (Experimental): Patients will be offered 4 courses of S-Gboxin during standard treatment. Each course (18 days) consists of twice daily intake of S-Gboxin for 14 days and four days of rest. Each dose of S-Gboxin is packed in a gelatin capsule with a bandage and applied markings.
  Interventions: Biological: S-Gboxin

INTERVENTIONS:
Biological: S-Gboxin — Gboxin specifically inhibits the growth of human glioblastoma cells but not normal cells. Gboxin rapidly and irreversibly impairs oxygen consumption in glioblastoma cells. Its positive charge for binding to mitochondrial oxidative phosphorylation complexes is dependent on the proton gradient of the inner mitochondrial membrane, and it inhibits F 0 F 1 ATP synthase activity in tumor cells. S-Gboxin crosses the blood-brain barrier at therapeutically effective concentrations.
  Other Names: oxidative phosphorylation inhibitor; OXPHOS inhibitor; suppression of oxidative phosphorylation

SUMMARY:
The objective of this pilot study is to evaluate the efficacy of adding S-Gboxin to standard RT/TMZ treatment protocols in patients with glioblastoma multiforme (GBM) or midline glioma (DMG), regardless of their mutation status

DETAILED DESCRIPTION:
This is a pilot study to evaluate the efficacy of adding the mitochondrial oxidative phosphorylation inhibitor S-Gboxin (OXPHOS) to standard treatment for glioblastoma multiforme or glioma.

Subjects will start oral S-gboxin orally twice daily and will evaluate the patients and vital status if they tolerate this dose at 3, 7and 15 days after initiation.

Patients will undergo MRI scans before treatment and then at multiple time points during their participation in this Clinical Trial to monitor early tumor response to treatment ( MRI dates will be scheduled by the clinical trial coordinator)

Peripheral blood samples will be collected at baseline, days 1-7-15-28-36-72 to compare biological indicators of treatment response. In some cases, circulating tumor cells (CTCs) will be monitored by real-time qRT-PCR to correlate with clinical data.

Patients will also be assessed for the side effects they experience. Disease-free and overall survival outcomes will be recorded.

Patients will also have their depressive symptoms, quality of life, and neurocognitive function assessed at multiple time points during and after treatment.

After completion of the study, patients will be followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Glioblastoma according to RANO criteria by contrast-enhanced MRI or PET-CT (including diffuse midline glioma, gliosarcoma or giant cell glioblastoma), relapse or disease progression
* patient is able to understand and give consent to participate in the study
* Karnofsky performance score ≥ 60
* women of childbearing potential must have a negative pregnancy test result no later than 7 days before registration

Exclusion Criteria:

* pregnant
* known allergies
* active treatment on annotner clinical trial
* inability to complete with protocol or studio procedures.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2027-10-10 (Estimated); Study Completion 2027-12-10 (Estimated)

PRIMARY OUTCOMES:
Brain tumor metabolism as measured by PET and MRI | Up to 6 month
  The standardized uptake value (SUV) of HGG will be measured. SUV is a standard PET measurement. MRI with contrast will evaluate the change in tumor size before and after therapy S-Gboxin

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 12 month
  Kaplan-Meier survival estimates for OS will be presented with using Greenwood's formula at 12 months.
Incidence of adverse events graded according to the Common Toxicity Criteria for Adverse Events (CTCAE) version (v)4.03 | Up to 1 month after last dose of S-Gboxin
  The data will be organized by major organ system and MedDRA severity after completion of the Clinical Study.

CONTACTS AND LOCATIONS:
Locations (3):
- Tbilisi Cancer Centre, Tbilisi, Georgia
- Kazakh Institute of Oncology and Radiology, Almaty, Kazakhstan
- National Cancer Institute, Kyiv, Ukraine

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF
Time Frame: documents will be available 3 months after completion of the research
Access Criteria: free access
URL: https://swissbio.zuerich/

REFERENCES:
- See also: Gboxin is an oxidative phosphorylation inhibitor that targets glioblastoma — https://pmc.ncbi.nlm.nih.gov/articles/PMC6655586/
- See also: Cancer cell-mitochondria hybrid membrane coated Gboxin loaded nanomedicines for glioblastoma treatment — https://www.nature.com/articles/s41467-023-40280-3
- See also: Nanomedicine and Immunotherapy for recurrent glioblastoma — https://braintumourresearch.org/blogs/research-campaigning-news/nanomedicine-and-immunotherapy-for-recurrent-glioblastoma?srsltid=AfmBOooU1XGjeuMxSBaBzWn4EGMFvsiNIktJRm4p7Ey8XVnJTor2oYHS